CLINICAL TRIAL: NCT00484289
Title: A Phase III, Multi-center, Open-label, Uncontrolled, Long-term Study to Evaluate the Safety of Abatacept (BMS-188667) in Japanese Subjects With Rheumatoid Arthritis Having Completed Clinical Studies IM101-071, IM101-034, and Also Special DMARD Failures
Brief Title: A Phase III Study of Abatacept in Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-129
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Participants from Phase I study (IM101-034) (Experimental)
  Interventions: Drug: Abatacept
- Arm 2: Participants from Phase II study (IM101-071) (Experimental)
  Interventions: Drug: Abatacept
- Arm 3: New Participants with Methotrexate (MTX) Intolerance (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Vials (250 mg/vial), Intravenous, Weight-tiered dose of abatacept (equivalent to 10 mg/kg) based on their body weight at the enrollment visit; 500 mg for participants < 60 kg, 750 mg for participants 60 to 100 kg and 1,000 mg for participants > 100 kg, administered over a period of approximately 30 minutes at week 0, 2, 4 and every 4 weeks thereafter, until approved in Japan and was continued as a post-marketing study until the completion of the shift to a commercially available product.
  Other Names: Orencia®; BMS-188667

SUMMARY:
The purpose of this study is to demonstrate the safety of chronic use of abatacept in Japanese Subjects with Rheumatoid Arthritis (RA) having completed clinical studies IM101-071, IM101-034, and also Disease Modifying Anti-Rheumatic Drugs (DMARDs) failures with MTX intolerance.

ELIGIBILITY:
Inclusion Criteria

* The participants who completed the 169 days, full study period of Phase II (IM101-071) and were not administered other biologics between completion of IM101-071 and registration of this long-term study.
* The participants of the Phase I study (IM101-034), who received abatacept, except participants who were withdrawn from the study due to safety problems related to abatacept.
* New subjects with MTX intolerance: rheumatoid arthritis (RA) patients to whom MTX cannot be administered for safety reasons and who present an inadequate response to disease-modifying antirheumatic drugs (DMARDs;excluding MTX) or biologics (new subjects with MTX intolerance: RA patients who present an inadequate response to DMARDs).

Exclusion Criteria

* Women of childbearing potential (WOCBP) who were unwilling or unable to use an acceptable method of contraception.
* Participants who have received non approved or investigational biologics (other than abatacept from previous or ongoing studies in Japan) at registration.
* Participants who have received treatment with any investigational drug within 56 days before registration or five half-lives (whichever is the longest).
* Participants currently receiving treatment with leflunomide, mycophenolate mofetil, calcineurine inhibitors such as cyclosporine and tacrolimus, D-Penicillamine, Cyclophosphamide, or immunoadsorption columns.
* The participants who completed Phase II (IM101-071) are not applicable in the following instances at time of registration: with active vasculitis, symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral disease, breast cancer, or a history of cancer within the last 5 years, evidence of active or latent bacterial , viral infections, any serious or chronic, at risk of tuberculosis (TB), with any opportunistic infections, laboratory values of hemoglobin < 8.5 g/dL, white blood cells (WBC) < 3,000/mm^3, Platelets < 100,000/mm^3, Serum creatinine > 2 times upper limit of normal (ULN), Serum alanine transaminase or aspartate aminotransferase > 2 times ULN.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- Japan (30):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Goshogawara-Shi, Aomori
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukui-shi, Fukui
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-Shi, Fukuoka
  - Local Institution, Higashi-Hiroshima-Shi, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanzaki-Gun, Hyōgo
  - Local Institution, Kato-Gun, Hyōgo
  - Local Institution, Hitachi-Shi, Ibaraki
  - Local Institution, Tsukuba, Ibaraki
  - Local Institution, Sagamihara-Shi, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nagano, Nagano
  - Local Institution, Tsukubo-Gun, Okayama-ken
  - Local Institution, Kawachinagano-Shi, Osaka
  - Local Institution, Ureshino-Shi, Saga-ken
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Kawagoe-Shi, Saitama
  - Local Institution, Kitamoto-Shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Kawachigun, Tochigi
  - Local Institution, Shimotsuke-Shi, Tochigi
  - Local Institution, Arakawa-Ku, Tokyo
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Setagaya-Ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Takaoka-Shi, Toyama
  - Local Institution, Chiba

REFERENCES:
- [Derived] Takeuchi T, Matsubara T, Urata Y, Suematsu E, Ohta S, Honjo S, Abe T, Yamamoto A, Miyasaka N; Japan Abatacept Study Group. Phase III, multicenter, open-label, long-term study of the safety of abatacept in Japanese patients with rheumatoid arthritis and an inadequate response to conventional or biologic disease-modifying antirheumatic drugs. Mod Rheumatol. 2014 Sep;24(5):744-53. doi: 10.3109/14397595.2014.899179. Epub 2014 Apr 23. PMID 24754273
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants From Phase I Study (IM101-034); Abatacept 10mg/kg: Participants with rheumatoid arthritis (RA) who participated in the phase I study (IM101-034). Weight-tiered dose of abatacept (equivalent to 10 mg/kg) based on their body weight at the enrollment visit was administered at Week 0, 2, 4 and every 4 weeks thereafter, as an intravenous (IV) infusion.
- Participants From Phase II Study(IM101-071); Abatacept 10mg/kg: Participants with RA who participated in the phase II study (IM101-071). Weight-tiered dose of abatacept (equivalent to 10 mg/kg) based on their body weight at the enrollment visit was administered at Week 0, 2, 4 and every 4 weeks thereafter, as an IV infusion.
- New Participants With MTX Intolerance; Abatacept 10 mg/kg: Participants with RA in whom methotrexate (MTX) could not be administered for safety reasons and who presented an inadequate response to disease-modifying antirheumatic drugs (DMARDs [excluding MTX]) and biologics. Weight-tiered dose of abatacept (equivalent to 10 mg/kg), based on their body weight at the enrollment visit, was administered at Week 0, 2, 4 and every 4 weeks thereafter, as an IV infusion.
Period: Long Term Phase
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Started | 13 | 178 | 26
Completed | 10 (Completed participants entered postmarketing phase.) | 142 (Completed participants entered postmarketing phase.) | 10 (Completed participants entered postmarketing phase.)
Not Completed | 3 | 36 | 16
Not completed — Adverse Event | 1 | 17 | 5
Not completed — Withdrawal by Subject | 0 | 7 | 6
Not completed — Inadequate response | 2 | 7 | 4
Not completed — Other Reason | 0 | 5 | 1
Period: Post Marketing Phase
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Started | 10 | 142 | 10
Completed | 10 | 141 | 10
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg | Total
Number analyzed (Participants) | 13 | 178 | 26 | 217
Age Continuous [Mean (Standard Deviation); unit: years] | 52.8 (11.6) | 53.2 (11.5) | 57.8 (10.6) | 53.8 (11.4)
Age, Customized [Number; unit: participants]
  20 - 29 years | 1 | 7 | 0 | 8
  30 - 39 years | 2 | 13 | 1 | 16
  40 - 49 years | 0 | 39 | 5 | 44
  50 - 59 years | 6 | 70 | 7 | 83
  ≥ 60 years | 4 | 49 | 13 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 146 | 19 | 177
  Male | 1 | 32 | 7 | 40
Weight [Mean (Standard Deviation); unit: kg] | 55.2 (9.7) | 56.9 (9.4) | 53.9 (10.8) | 56.5 (9.6)
Duration of Rheumatoid Arthritis [Number; unit: participants]
  <= 2 years | 0 (9.0) | 24 (7.3) | 2 (10.1) | 26 (7.9)
  >2 to <= 5 years | 2 | 45 | 4 | 51
  > 5 to <= 10 years | 2 | 57 | 12 | 71
  > 10 years | 9 | 52 | 8 | 69
American College of Rheumatology (ACR) Functional Status Classification [Number; unit: participants] — ACR Classification Criteria for Determining Progression of Rheumatoid Arthritis - Class I: Completely able to perform usual activities of daily living; II: Able to perform usual self-care and vocational activities, but limited in avocational activities ; III: Able to perform usual self-care activities, but limited in vocational and avocational activities ; IV: Limited ability to perform usual self-care, vocational, and avocational activities
  participants
    Class I | 0 | 29 | 0 | 29
    Class II | 12 | 112 | 17 | 141
    Class III | 1 | 37 | 9 | 47
    Class IV | 0 | 0 | 0 | 0
Number of Tender Joints [Mean (Standard Deviation); unit: joints] — Tender joints are an indicator of Rheumatoid Arthritis. The number of tender joints in a standard 68 joint count was evaluated. The number of tender joints ranges from 0 tender joints to 68, where an increased number of tender joints indicates increasing level of disease severity.
  joints | 8.4 (5.2) | 14.3 (11.2) | 22.7 (13.3) | 14.9 (11.6)
Number of Swollen Joints [Mean (Standard Deviation); unit: joints] — Swollen joints are an indicator of Rheumatoid Arthritis. The number of swollen joints in a standard 66 joint count was evaluated. The number of swollen joints ranges from 0 swollen joints to 66, where an increased number of swollen joints indicate increasing level of disease severity.
  joints | 9.1 (4.7) | 11.6 (8.7) | 17.2 (10.0) | 12.1 (8.9)
Participant Pain Assessment [Mean (Standard Deviation); unit: units on a scale] — The participant self-reported pain assessment is a core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale (VAS) with 0 mm representing "no pain" and 100 mm representing the "most pain possible".
  units on a scale | 43.1 (23.5) | 52.3 (24.9) | 80.6 (20.1) | 55.1 (26.0)
Physical Function (Health Assessment Questionnaire [HAQ]) [Mean (Standard Deviation); unit: units on a scale] — The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ disability Index.
  units on a scale | 0.98 (0.57) | 1.16 (0.75) | 1.80 (0.90) | 1.22 (0.79)
Physician Global Assessment [Mean (Standard Deviation); unit: Units on a scale] — Physician Global Assessment of the participant's disease activity using a visual analog scale (VAS) of 0 - 100 mm with 100 mm being the worst case), a component of the ACR criteria.
  Units on a scale | 56.5 (24.7) | 47.5 (24.0) | 75.5 (16.5) | 51.4 (24.9)
Participant Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Participants used a horizontal visual analog scale (VAS) of 100 mm for overall assessment of rheumatoid arthritis. Scale ranged from 0 (very well) to 100 (very poor). Participants were instructed to draw a vertical through a horizontal line to indicate state of rheumatoid arthritis. Distance from the "very well" end of the horizontal line to the vertical line drawn by the participant was the global disease assessment score on a scale of 1-10, where 1=controlled or equivocal rheumatoid arthritis activity, 1.1-4=mild activity, 4.1-8=moderate activity, and 8.1-10=high activity.
  units on a scale | 47.1 (20.7) | 50.8 (23.8) | 77.3 (20.4) | 53.7 (24.8)
C-Reactive Protein (CRP) Level [Mean (Standard Deviation); unit: mg/dL] — CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of CRP can be used to determine DAS 28.
  mg/dL | 1.84 (2.84) | 2.32 (2.18) | 4.67 (3.65) | 2.57 (2.55)
Morning stiffness [Mean (Standard Deviation); unit: minutes] | 117.7 (201.3) | 72.7 (124.9) | 166.6 (195.7) | 86.7 (143.0)
Rheumatoid Factor Status [Number; unit: participants] — Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which in itself is an antibody. RF and IgG join to form immune complexes which contribute to the disease process. RF levels are considered positive if value is >20 IU/mL and considered negative if value is <20.
  participants
    Negative (<=20 IU/mL) | 1 | 24 | 4 | 29
    Positive (>20 IU/mL) | 12 | 154 | 22 | 188
Methotrexate Usage at Registration [Mean (Standard Deviation); unit: mg/week] — n=9, 175, and 0 for participants from phase I study,phase II study, and new participants with MTX, respectively.
  mg/week | 7.11 (1.45) | 7.11 (1.07) | NA (NA) — This arm had only participants to whom MTX could not be administered for safety reasons | 7.11 (1.09)
Oral Corticosteroids Usage at Registration [Mean (Standard Deviation); unit: mg/day] — Dosage of oral corticosteroids was calculated using prednisolone volume. n=13, 146, and 23 for participants from phase I study, phase II study, and new participants with MTX, respectively.
  mg/day | 6.15 (2.37) | 5.67 (2.38) | 6.78 (2.48) | 5.85 (2.41)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE), and Discontinuations Due to AEs
Description: AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event. Both subjective and objective AEs and SAEs are included.
Time Frame: From initiation of the study drug (31 Mar 2008) to data cutoff (27 Dec 2010). The overall mean duration of exposure to the study drug was approximately 3 years (34.3 ± 10.7 months).
Population: All treated participants who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  SAEs | 4 | 50 | 14
  Drug-related SAEs | 2 | 26 | 9
  AEs | 13 | 176 | 24
  Drug-related AEs | 13 | 165 | 24
  Discontinuation due to SAEs | 0 | 14 | 5
  Discontinuation due to AEs | 1 | 18 | 5
  Deaths | 0 | 1 | 0

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR 20) Response Over Time
Description: ACR 20 response requires a participant to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease activity, participant global assessment of disease activity, participant global assessment of pain, C-reactive protein, and degree of disability in Health Assessment Questionnaire score.
Time Frame: At weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192.
Population: All treated participants who received at least 1 dose of the study drug. n = number of participants assessed at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
percentage of participants
  Week 4; (n=13, 178,26) | 30.8 [9.1 to 61.4] | 29.2 [22.7 to 36.5] | 34.6 [17.2 to 55.7]
  Week 12; (n=13, 178,24) | 76.9 [46.2 to 95.0] | 47.2 [39.7 to 54.8] | 58.3 [36.6 to 77.9]
  Week 24; (n=13, 176, 23) | 76.9 [46.2 to 95.0] | 59.7 [52.0 to 67.0] | 78.3 [56.3 to 92.5]
  Week 36; (n=13, 175, 20) | 69.2 [38.6 to 90.9] | 61.7 [54.1 to 68.9] | 90.0 [68.3 to 98.8]
  Week 48; (n=13, 170, 18) | 61.5 [31.6 to 86.1] | 63.5 [55.8 to 70.8] | 88.9 [65.3 to 98.6]
  Week 60; (n=13, 165, 17) | 69.2 [38.6 to 90.9] | 69.7 [62.1 to 76.6] | 94.1 [71.3 to 99.9]
  Week 72; (n=13, 161, 17) | 84.6 [54.6 to 98.1] | 67.7 [59.9 to 74.8] | 94.1 [71.3 to 99.9]
  Week 84; (n=13, 161, 17) | 61.5 [31.6 to 86.1] | 67.1 [59.2 to 74.3] | 100.0 [80.5 to 100.0]
  Week 96; (n=13, 160, 17) | 69.2 [38.6 to 90.9] | 63.8 [55.8 to 71.2] | 82.4 [56.6 to 96.2]
  Week 108; (n=13, 156, 15) | 53.8 [25.1 to 80.8] | 67.9 [60.0 to 75.2] | 100.0 [78.2 to 100.0]
  Week 120; (n=13, 154, 15) | 69.2 [38.6 to 90.9] | 69.5 [61.6 to 76.6] | 100.0 [78.2 to 100.0]
  Week 132; (n=13, 151, 14) | 61.5 [31.6 to 86.1] | 68.9 [60.8 to 76.2] | 100.0 [76.8 to 100.0]
  Week 144; (n=12, 142, 13) | 58.3 [27.7 to 84.8] | 69.7 [61.5 to 77.1] | 84.6 [54.6 to 98.1]
  Week 156; (n=11, 113, 12) | 63.6 [30.8 to 89.1] | 66.4 [56.9 to 75.0] | 100.0 [73.5 to 100.0]
  Week 168; (n=10, 80, 8) | 80.0 [44.4 to 97.5] | 71.3 [60.0 to 80.8] | 100.0 [63.1 to 100.0]
  Week 180; (n=8, 56, 4) | 62.5 [24.5 to 91.5] | 69.6 [55.9 to 81.2] | 100.0 [39.8 to 100.0]
  Week 192; (n=3, 7, 1) | 66.7 [9.4 to 99.2] | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0]

3. Secondary Outcome: Percentage of Participants With ACR 50 Response Over Time
Description: ACR 50 response requires a participant to have a 50% reduction in the number of swollen and tender joints, and a reduction of 50% in three of the following five parameters: physician global assessment of disease activity, participant global assessment of disease activity, participant global assessment of pain, C-reactive protein, and degree of disability in Health Assessment Questionnaire score.
Time Frame: At weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
percentage of participants
  Week 4; (n=13, 178, 26) | 15.4 [1.9 to 45.4] | 6.2 [3.1 to 10.8] | 0 [0 to 13.2]
  Week 12; (n=13, 178,24) | 38.5 [13.9 to 68.4] | 16.3 [11.2 to 22.6] | 29.2 [12.6 to 51.1]
  Week 24; (n=13, 176, 23) | 30.8 [9.1 to 61.4] | 25.6 [19.3 to 32.7] | 47.8 [26.8 to 69.4]
  Week 36; (n=13, 175, 20) | 38.5 [13.9 to 68.4] | 28.6 [22.0 to 35.9] | 50.0 [27.2 to 72.8]
  Week 48; (n=13, 170, 18) | 15.4 [1.9 to 45.4] | 38.8 [31.5 to 46.6] | 72.2 [46.5 to 90.3]
  Week 60; (n=13, 165, 17) | 30.8 [9.1 to 61.4] | 42.4 [34.8 to 50.3] | 58.8 [32.9 to 81.6]
  Week 72; (n=13, 161, 17) | 46.2 [19.2 to 74.9] | 43.5 [35.7 to 51.5] | 70.6 [44.0 to 89.7]
  Week 84; (n=13, 161, 17) | 38.5 [13.9 to 68.4] | 42.2 [34.5 to 50.3] | 70.6 [44.0 to 89.7]
  Week 96; (n=13, 160, 17) | 23.1 [5.0 to 53.8] | 38.1 [30.6 to 46.1] | 58.8 [32.9 to 81.6]
  Week 108; (n=13, 156, 15) | 23.1 [5.0 to 53.8] | 42.3 [34.4 to 50.5] | 66.7 [38.4 to 88.2]
  Week 120; (n=13, 154, 15) | 46.2 [19.2 to 74.9] | 45.5 [37.4 to 53.7] | 93.3 [68.1 to 99.8]
  Week 132; (n=13, 151, 14) | 38.5 [13.9 to 68.4] | 43.7 [35.7 to 52.0] | 85.7 [57.2 to 98.2]
  Week 144; (n=12, 142, 13) | 25.0 [5.5 to 57.2] | 47.2 [38.8 to 55.7] | 69.2 [38.6 to 90.9]
  Week 156; (n=11, 113, 12) | 36.4 [10.9 to 69.2] | 47.8 [38.3 to 57.4] | 83.3 [51.6 to 97.9]
  Week 168; (n=10, 80, 8) | 30.0 [6.7 to 65.2] | 47.5 [36.2 to 59.0] | 87.5 [47.3 to 99.7]
  Week 180; (n=8, 56, 4) | 12.5 [0.3 to 52.7] | 51.8 [38.0 to 65.3] | 75.0 [19.4 to 99.4]
  Week 192; (n=3, 7, 1) | 66.7 [9.4 to 99.2] | 71.4 [29.0 to 96.3] | 100.0 [2.5 to 100.0]

4. Secondary Outcome: Percentage of Participants With ACR 70 Response Over Time
Description: ACR 70 response requires a participant to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in three of the following five parameters: physician global assessment of disease activity, participant global assessment of disease activity, participant global assessment of pain, C-reactive protein, and degree of disability in Health Assessment Questionnaire score.
Time Frame: At weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, and 192.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
percentage of participants
  Week 4; (n=13, 178, 26) | 7.7 [0.2 to 36.0] | 0 [0 to 2.1] | 0 [0 to 13.2]
  Week 12; (n=13, 178, 24) | 7.7 [0.2 to 36.0] | 5.6 [2.7 to 10.1] | 8.3 [1.0 to 27.0]
  Week 24; (n=13, 176, 23) | 7.7 [0.2 to 36.0] | 10.8 [6.6 to 16.3] | 21.7 [7.5 to 43.7]
  Week 36; (n=13, 175, 20) | 15.4 [1.9 to 45.4] | 11.4 [7.1 to 17.1] | 20.0 [5.7 to 43.7]
  Week 48; (n=13, 170, 18) | 15.4 [1.9 to 45.4] | 15.3 [10.2 to 21.6] | 27.8 [9.7 to 53.5]
  Week 60; (n=13, 165, 17) | 15.4 [1.9 to 45.4] | 19.4 [13.7 to 26.3] | 29.4 [10.3 to 56.0]
  Week 72; (n=13, 161, 17) | 15.4 [1.9 to 45.4] | 18.6 [12.9 to 25.5] | 23.5 [6.8 to 49.9]
  Week 84; (n=13, 161, 17) | 7.7 [0.2 to 36.0] | 17.4 [11.9 to 24.1] | 23.5 [6.8 to 49.9]
  Week 96; (n=13, 160, 17) | 7.7 [0.2 to 36.0] | 19.4 [13.6 to 26.4] | 23.5 [6.8 to 49.9]
  Week 108; (n=13, 156, 15) | 7.7 [0.2 to 36.0] | 15.4 [10.1 to 22.0] | 33.3 [11.8 to 61.6]
  Week 120; (n=13, 154, 15) | 7.7 [0.2 to 36.0] | 19.5 [13.5 to 26.6] | 46.7 [21.3 to 73.4]
  Week 132; (n=13, 151, 14) | 0 [0 to 24.7] | 20.5 [14.4 to 27.9] | 42.9 [17.7 to 71.1]
  Week 144; (n=12, 142, 13) | 0 [0 to 26.5] | 21.8 [15.3 to 29.5] | 23.1 [5.0 to 53.8]
  Week 156; (n=11, 113, 12) | 0 [0 to 28.5] | 25.7 [17.9 to 34.7] | 33.3 [9.9 to 65.1]
  Week 168; (n=10, 80, 8) | 0 [0 to 30.8] | 27.5 [18.1 to 38.6] | 62.5 [24.5 to 91.5]
  Week 180; (n=8, 56, 4) | 0 [0 to 36.9] | 33.9 [21.8 to 47.8] | 50.0 [6.8 to 93.2]
  Week 192; (n=3, 7, 1) | 0 [0 to 70.8] | 14.3 [0.4 to 57.9] | 100.0 [2.5 to 100.0]

5. Secondary Outcome: Baseline (BL) and Postbaseline (PBL) Disease Activity Scores (DAS 28)
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale of 100 mm. The DAS28 has numeric thresholds that define high disease activity (change of > 5.1), low disease activity (change of ≤ 3.2) and remission (< 2.6). Please see outcome 8 for change from BL data.
Time Frame: At BL (week 0), week 24, 48, 96, 144, and 192.
Population: All treated participants who received at least 1 dose of the study drug. n = participants with both BL and PBL measurement at a given time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24- BL (n=13, 176, 21) | 4.4 (1.0) | 4.8 (1.4) | 6.3 (1.0)
  Week 24- PBL (n=13, 176, 21) | 3.0 (1.1) | 3.2 (1.1) | 4.0 (1.9)
  Week 48- BL (n=13, 168, 18) | 4.4 (1.0) | 4.8 (1.4) | 6.3 (1.0)
  Week 48- PBL (n=13, 168, 18) | 3.0 (1.1) | 2.9 (1.1) | 3.5 (1.4)
  Week 96- BL (n=13, 159, 17) | 4.4 (1.0) | 4.8 (1.4) | 6.2 (1.0)
  Week 96- PBL (n=13, 159, 17) | 3.3 (1.0) | 2.8 (1.0) | 3.2 (1.0)
  Week 144- BL (n=12, 142, 13) | 4.3 (0.9) | 4.9 (1.4) | 6.3 (1.0)
  Week 144- PBL (n=12, 142, 13) | 3.0 (0.9) | 2.8 (1.0) | 3.2 (1.2)
  Week 192- BL (n=3, 7, 1) | 4.6 (1.6) | 5.4 (0.9) | 7.9 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.
  Week 192- PBL (n=3, 7, 1) | 2.6 (1.2) | 3.1 (1.4) | 1.9 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.

6. Secondary Outcome: Change From Baseline in DAS 28 Scores at Week 24, 48, 96, 144, and 192
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale of 100 mm. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (≤ 3.2) and remission (< 2.6). Please refer to outcome 7 for BL and PBL values.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24 (n=13, 176, 21) | -1.4 [-2.0 to -0.8] | -1.7 [-1.8 to -1.5] | -2.3 [-2.9 to -1.7]
  Week 48 (n=13, 168, 18) | -1.4 [-2.0 to -0.9] | -1.9 [-2.1 to -1.7] | -2.8 [-3.3 to -2.3]
  Week 96 (n=13, 159, 17) | -1.1 [-1.7 to -0.6] | -2.0 [-2.3 to -1.8] | -3.0 [-3.6 to -2.4]
  Week 144 (n=12, 142, 13) | -1.3 [-1.8 to -0.8] | -2.1 [-2.3 to -1.9] | -3.1 [-4.0 to -2.2]
  Week 192 (n=3, 7, 1) | -2.0 [-3.4 to -0.6] | -2.3 [-3.6 to -1.1] | -6.0 [NA to NA] — Not applicable as there was only 1 participant in the group with both BL and PBL values.

7. Secondary Outcome: Number of Participants With DAS 28 Score Change ≥ 1.2 From Baseline at Weeks 24, 48, 96, 144, and 192
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale.
  Participants with DAS 28 score change ≥ 1.2 from BL were considered to have improvement.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Week 24 (n=13, 176, 21) | 9 | 113 | 17
  Week 48 (n=13, 168, 18) | 8 | 114 | 16
  Week 96 (n=13, 159, 17) | 7 | 111 | 16
  Week 144 (n=12, 142, 13) | 6 | 107 | 12
  Week 192 (n=3, 7, 1) | 3 | 5 | 1

8. Primary Outcome: Number of Participants With Abnormal Laboratory Changes (ALC)
Description: The laboratory tests were analyses included enzyme, gastrointestinal, hematology, hepatobiliary, lipid, metabolic, nutritional, blood gas, microbiology, serology, protein, chemistry, renal, urinary tract, urinalyses, water, electrolyte and mineral investigations.
Time Frame: as for outcome 1
Population: All treated participants who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Participants with Serious ALC | 0 | 0 | 1
  Discontinuations due Serious ALC | 0 | 0 | 0
  Participants with drug related Serious ALC | 0 | 0 | 1
  Participants with ALC | 0 | 1 | 0
  Discontinuations due ALC | 7 | 125 | 19
  Discontinuations due ALC | 6 | 102 | 13

9. Secondary Outcome: Number of Participants With Low Disease Activity Score (DAS 28 Score ≤ 3.2) at Weeks 24, 48, 96, 144, 192
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale. Participants with DAS 28 score ≤ 3.2 were considered to have low disease activity.
Time Frame: At weeks 24, 48, 96, 144, and 192.
Population: All treated participants who received at least 1 dose of the study drug. n = participants with available scores at the given time point.
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Week 24 (n=13, 176, 21) | 9 | 95 | 6
  Week 48 (n=13, 168, 18) | 9 | 105 | 7
  Week 96 (n=13, 159, 17) | 6 | 101 | 6
  Week 144 (n=12, 142, 13) | 6 | 95 | 7
  Week 192 (n=3, 7, 1) | 2 | 3 | 1

10. Secondary Outcome: Number of Participants in Remission (DAS 28 Score < 2.6) at Weeks 24, 48, 96, 144, 192
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale.
  Participants with DAS 28 score < 2.6 were considered to be in remission.
Time Frame: At weeks 24, 48, 96, 144, and 192.
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Week 24 (n=13, 176, 21) | 6 | 60 | 6
  Week 48 (n=13, 168, 18) | 4 | 75 | 5
  Week 96 (n=13, 159, 17) | 3 | 75 | 5
  Week 144 (n=12, 142, 13) | 4 | 71 | 3
  Week 192 (n=3, 7, 1) | 2 | 2 | 1

11. Secondary Outcome: Percentage of Participants Who Achieved a Reduction of At Least 0.3 Units From Baseline in Health Assessment Questionnaire (HAQ) at Weeks 24, 48, 96, 144, 192
Description: The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from BL in HAQ.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
percentage of participants
  Week 24 (n=13, 176, 23) | 38.5 [13.9 to 68.4] | 39.2 [31.9 to 46.8] | 52.2 [30.6 to 73.2]
  Week 48 (n=13, 170, 18) | 30.8 [9.1 to 61.4] | 41.2 [33.7 to 49.0] | 77.8 [52.4 to 93.6]
  Week 96 (n=13, 160, 17) | 46.2 [19.2 to 74.9] | 47.5 [39.6 to 55.5] | 76.5 [50.1 to 93.2]
  Week 144 (n=12, 142, 13) | 50.0 [21.1 to 78.9] | 48.6 [40.1 to 57.1] | 69.2 [38.6 to 90.9]
  Week 192 (n=3, 7, 1) | 100.0 [29.2 to 100.0] | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0]

12. Secondary Outcome: Baseline and Postbaseline Physical Component Summary (PCS) of Health-Related Quality of Life (SF-36) Scores
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role functioning [physical], bodily pain, and general health) and 4 mental subscales (vitality, social function, role emotional, and mental health). All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful.Please see outcome 14 for change from BL data.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: All treated participants who received at least 1 dose of the study drug. n = participants with both BL and PBL measurement at a given point time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24- BL (n=13, 176, 23) | 34.2 (14.5) | 30.3 (15.2) | 19.0 (12.5)
  Week 24- PBL (n=13, 176, 23) | 40.6 (12.6) | 38.5 (14.3) | 30.3 (17.1)
  Week 48- BL (n=13, 170, 18) | 34.2 (14.5) | 30.4 (15.2) | 20.1 (12.4)
  Week 48- PBL (n=13, 170, 18) | 40.9 (11.1) | 40.1 (13.7) | 37.1 (14.0)
  Week 96- BL (n=13, 160, 17) | 34.2 (14.5) | 29.8 (15.2) | 19.9 (12.7)
  Week 96- PBL (n=13, 160, 17) | 38.7 (12.6) | 40.3 (13.2) | 37.5 (13.5)
  Week 144- BL (n=12, 142, 13) | 32.9 (14.4) | 30.6 (15.1) | 21.1 (14.0)
  Week 144- PBL (n=12, 142, 13) | 37.8 (14.5) | 39.2 (13.7) | 32.9 (14.2)
  Week 192- BL (n=3, 7, 1) | 24.6 (10.9) | 22.8 (12.2) | 12.5 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.
  Week 192- PBL (n=3, 7, 1) | 30.4 (24.8) | 38.5 (16.1) | 37.0 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.

13. Secondary Outcome: Change From Baseline in Physical Component Summary (PCS) of Health-Related Quality of Life (SF-36) Score at Weeks 24, 48, 96, 144, and 192
Description: The SF-36 covers 8 health dimensions including 4 physical (physical function, role functioning [physical], bodily pain, and general health) and 4 mental subscales (vitality, social function, role emotional, and mental health). All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from a minimum of 0 to a maximum of 100, higher score indicating better quality of life. Improvements of >3 points were considered clinically meaningful. Please see outcome 13 for BL and PBL values.
Time Frame: At baseline (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24 (n=13, 176, 23) | 6.5 [0 to 13.0] | 8.2 [6.4 to 10.0] | 11.3 [5.2 to 17.5]
  Week 48 (n=13, 170, 18) | 6.7 [0.3 to 13.1] | 9.7 [7.7 to 11.7] | 17.1 [11.1 to 23.0]
  Week 96 (n=13, 160, 17) | 4.5 [-4.5 to 13.6] | 10.4 [8.5 to 12.4] | 17.6 [9.7 to 25.5]
  Week 144 (n=12, 142, 13) | 4.8 [-5.3 to 14.9] | 8.6 [6.6 to 10.6] | 11.8 [4.4 to 19.1]
  Week 192 (n=3, 7, 1) | 5.7 [-79.9 to 91.4] | 15.7 [0.7 to 30.8] | 24.6 [NA to NA] — Not applicable as there was only 1 participant in the group with both BL and PBL values.

14. Secondary Outcome: Baseline and Postbaseline Mental Component Summary (MCS) of Health-Related Quality of Life (SF-36) Scores
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role functioning [physical], bodily pain, and general health) and 4 mental subscales (vitality, social function, role emotional, and mental health). All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful. Please see outcome 14 for change from BL data.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24- BL (n=13, 176, 23) | 41.6 (12.4) | 48.6 (8.5) | 41.7 (9.8)
  Week 24- PBL (n=13, 176, 23) | 45.2 (8.9) | 51.2 (7.5) | 49.5 (10.5)
  Week 48- BL (n=13, 170, 18) | 41.6 (12.4) | 48.6 (8.5) | 43.2 (9.6)
  Week 48- PBL (n=13, 170, 18) | 49.0 (8.0) | 51.6 (8.1) | 49.9 (7.5)
  Week 96- BL (n=13, 160, 17) | 41.6 (12.4) | 48.6 (8.5) | 43.6 (9.8)
  Week 96- PBL (n=13, 160, 17) | 49.9 (7.2) | 50.6 (7.5) | 51.6 (8.2)
  Week 144- BL (n=12, 142, 13) | 41.6 (13.0) | 48.5 (8.6) | 42.2 (9.4)
  Week 144- PBL (n=12, 142, 13) | 51.1 (7.6) | 50.6 (7.3) | 51.1 (8.4)
  Week 192- BL (n=3, 7, 1) | 45.7 (20.4) | 45.4 (8.1) | 37.1 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.
  Week 192- PBL (n=3, 7, 1) | 60.7 (6.1) | 52.4 (12.5) | 69.3 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.

15. Secondary Outcome: Change From Baseline in Mental Component Summary (MCS) of Health-Related Quality of Life (SF-36) Score at Weeks 24, 48, 96, 144, and 192
Description: The SF-36 covers 8 health dimensions including 4 physical (physical function, role functioning [physical], bodily pain, and general health) and 4 mental subscales (vitality, social function, role emotional, and mental health). All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from a minimum of 0 to a maximum of 100, higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful.Please see outcome 15 for BL and PBL values.
Time Frame: At BL (Week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
Units on a Scale
  Week 24 (n=13, 176, 23) | 3.6 [-1.3 to 8.6] | 2.6 [1.5 to 3.7] | 7.7 [1.7 to 13.8]
  Week 48 (n=13, 170, 18) | 7.4 [2.5 to 12.3] | 3.0 [1.7 to 4.3] | 6.7 [1.4 to 11.9]
  Week 96 (n=13, 160, 17) | 8.3 [2.0 to 14.6] | 2.1 [0.7 to 3.4] | 8.0 [1.9 to 14.2]
  Week 144 (n=12, 142, 13) | 9.5 [3.4 to 15.6] | 2.1 [0.8 to 3.5] | 8.9 [1.9 to 15.9]
  Week 192 (n=3, 7, 1) | 15.0 [-49.5 to 79.6] | 7.0 [-5.2 to 19.3] | 32.1 [NA to NA] — Not applicable as there was only 1 participant in the group with both BL and PBL values.

16. Secondary Outcome: Baseline and Postbaseline C-reactive Protein (CRP) Levels
Description: CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA) and is a core component of the ACR scoring system. CRP was evaluated from serum samples. Increasing levels indicate increasing level of disease. Please see outcome 18 for change from BL data.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: All treated participants who received at least 1 dose of the study drug. n = number of participants with both BL and PBL measurement at a given point time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
mg/dL
  Week 24- BL (n=13, 176, 21) | 1.8 (2.8) | 2.3 (2.2) | 3.9 (3.1)
  Week 24- PBL (n=13, 176, 21) | 0.7 (0.7) | 0.8 (1.3) | 1.9 (2.5)
  Week 48- BL (n=13, 168, 18) | 1.8 (2.8) | 2.2 (2.1) | 4.1 (3.1)
  Week 48- PBL (n=13, 168, 18) | 1.1 (2.1) | 0.6 (1.1) | 0.9 (1.3)
  Week 96- BL (n=13, 159, 17) | 1.8 (2.8) | 2.3 (2.2) | 4.1 (3.2)
  Week 96- PBL (n=13, 159, 17) | 0.9 (1.3) | 0.5 (0.9) | 1.0 (1.0)
  Week 144- BL (n=12, 142, 13) | 1.9 (2.9) | 2.4 (2.2) | 4.2 (3.4)
  Week 144- PBL (n=12, 142, 13) | 1.2 (1.4) | 0.6 (1.5) | 0.6 (0.6)
  Week 192- BL (n=3, 7, 1) | 4.6 (5.4) | 1.7 (1.2) | 8.4 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.
  Week 192- PBL (n=3, 7, 1) | 1.4 (1.7) | 0.8 (1.6) | 0.2 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.

17. Secondary Outcome: Percentage Decrease in C-reactive Protein Levels From Baseline at Weeks 24, 48, 96, 144, and 192
Description: CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA) and is a core component of the ACR scoring system. CRP was evaluated from serum samples. Increasing levels indicate increasing level of disease, negative values indicate improvement. Percentage improvement from BL = (BL - PBL value) / BL value * 100. Please refer to outcome 17 for BL and PBL values.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
percentage improvement
  Week 24 (n=13, 176, 21) | -18.4 [-147.8 to 111.1] | 30.5 [-0.4 to 61.4] | 60.2 [42.7 to 77.7]
  Week 48 (n=13, 168, 18) | 12.0 [-35.9 to 59.9] | 31.9 [8.7 to 55.1] | 77.8 [65.2 to 90.3]
  Week 96 (n=13, 159, 17) | -3.3 [-77.9 to 71.3] | 40.5 [21.8 to 59.1] | 70.1 [51.0 to 89.2]
  Week 144 (n=12, 142, 13) | -71.9 [-188.7 to 44.9] | -39.3 [-191.5 to 113.0] | 79.9 [68.0 to 91.7]
  Week 192 (n=3, 7, 1) | 67.9 [52.0 to 83.7] | 39.7 [-83.2 to 162.6] | 97.4 [NA to NA] — Not applicable as there was only 1 participant in the group with both baseline and postbaseline values.

18. Secondary Outcome: Baseline and Postbaseline Rheumatoid Factor Levels
Description: Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. RF levels are considered positive if value is >20 and considered negative if value is <20. Please see outcome 20 for change from BL data.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
IU/mL
  Week 24- BL (n=13, 176, 21) | 200.2 (343.8) | 214.3 (383.3) | 630.8 (873.4)
  Week 24- PBL (n=13, 176, 21) | 127.5 (191.6) | 141.0 (289.2) | 573.9 (897.2)
  Week 48- BL (n=13, 168, 18) | 200.2 (343.8) | 217.3 (389.7) | 560.9 (893.0)
  Week 48- PBL (n=13, 168, 18) | 139.9 (241.8) | 149.5 (288.4) | 288.3 (482.8)
  Week 96- BL (n=13, 159, 17) | 200.2 (343.8) | 215.9 (393.9) | 590.9 (911.1)
  Week 96- PBL (n=13, 159, 17) | 186.9 (339.4) | 151.0 (285.8) | 216.8 (329.2)
  Week 144- BL (n=12, 142, 13) | 205.6 (358.5) | 229.0 (412.6) | 639.4 (990.8)
  Week 144- PBL (n=12, 142, 13) | 211.3 (359.8) | 173.7 (360.8) | 361.6 (663.9)
  Week 192- BL (n=3, 7, 1) | 314.3 (455.3) | 253.7 (307.6) | 2800.0 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.
  Week 192- PBL (n=3, 7, 1) | 315.0 (307.0) | 348.4 (521.6) | 197.0 (NA) — Not applicable as there was only 1 participant in the group with both BL and PBL values.

19. Secondary Outcome: Change From Baseline in Rheumatoid Factor Levels at Weeks 24, 48, 96, 144, and 192
Description: RF is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. RF levels are considered positive if value is >20 and considered negative if value is <20. Please refer to outcome 19 for BL and PBL values.
Time Frame: At BL (week 0), weeks 24, 48, 96, 144, and 192.
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
IU/mL
  Week 24 (n=13, 176, 21) | -72.6 [-197.5 to 52.2] | -73.2 [-102.8 to -43.7] | -56.9 [-149.5 to 35.7]
  Week 48 (n=13, 168, 18) | -60.2 [-137.9 to 17.4] | -67.8 [-100.4 to -35.2] | -272.6 [-494.0 to -51.2]
  Week 96 (n=13, 159, 17) | -13.2 [-63.3 to 36.8] | -64.9 [-103.3 to -26.6] | -374.1 [-704.9 to -43.2]
  Week 144 (n=12, 142, 13) | 5.7 [-43.0 to 54.4] | -55.3 [-97.2 to -13.3] | -277.8 [-708.2 to 152.7]
  Week 192 (n=3, 7, 1) | 0.7 [-471.3 to 472.7] | 94.7 [-122.5 to 311.9] | -2603 [NA to NA] — Not applicable as there was only 1 participant with both BL and BL measurements.

20. Secondary Outcome: Number of Participants Who Were Positive for Anti-abatacept and Anti-CTLA4-T Antibodies
Description: Validated enzyme-linked immunoassay (ELISA) method was used to measure anti-abatacept and anti-CTLA4-T antibody levels. For anti-abatacept antibody ELISA, a sample was considered seropositive if it had a titer of 400 or greater and if immunodepletion was observed. The responses that were negative in initial screen were reported as seronegative with a value of < 400. A sample was considered positive in CTLA4-T antibody ELISA if it had a titer of 25 or greater and if immunodepletion was observed.
Time Frame: At BL (week 0), weeks 24, 48, 72, 96, 120, 144, 168, and 192.
Population: All participants who received study treatment, and had BL and at least one PBL measurement for immunogenicity.
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Positive for anti-abatacept antibody | 2 | 19 | 2
  Positive for anti-CTLA4-T antibody | 0 | 19 | 1

21. Secondary Outcome: Abatacept PK Parameter: Total Body Clearance
Description: Total body clearance is the rate and extent at which the drug is eliminated from the body. The clearance of a drug is used to understand the processes involved in drug elimination, distribution and metabolism.
Time Frame: Samples were collected predose at week 8, 12, 16, 24; end of infusion at week 12; and at week 13-15 visits.
Population: All participants who received abatacept and had blood samples for assay.
Measure: Median (Full Range); unit: L/day
Groups:
- All Participants From IM101-129 Study: Participants with rheumatoid arthritis (RA) who participated in studies IM101-034 and IM101-071. Weight-tiered dose of abatacept (equivalent to 10 mg/kg) based on their body weight at the enrollment visit was administered at Weeks 0, 2, 4 and every 4 weeks thereafter, as an intravenous (IV) infusion.
Arm/Group | All Participants From IM101-129 Study
Number analyzed (Participants) | 113
L/day | 0.306 (0.098) [0.149 to 0.668]

22. Secondary Outcome: Abatacept PK Parameter: Area Under the Serum Concentration-time Curve at Steady State
Description: Area under the plasma concentration-time curve (AUCss) at steady state for each dosing interval was determined using the linear trapezoidal rule.
Time Frame: Samples were collected predose at week 8, 12, 16, 24; end of infusion at week 12; and at week 13-15 visits.
Population: All participants who received abatacept and had blood samples for assay.
Measure: Median (Full Range); unit: µg*h/mL
Arm/Group | All Participants From IM101-129 Study
Number analyzed (Participants) | 113
µg*h/mL | 42959.94 (12763.45) [17971.87 to 80321.29]

23. Secondary Outcome: Abatacept PK Parameter: Maximum Serum Concentration at Steady State
Description: Maximum plasma concentration is the maximum observed serum drug concentration at steady state (Css max).
Time Frame: Samples were collected predose at week 8, 12, 16, 24; end of infusion at week 12; and at week 13-15 visits.
Population: All participants who received abatacept and had blood samples for assay.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | All Participants From IM101-129 Study
Number analyzed (Participants) | 113
µg/mL | 241.62 (73.96) [68.15 to 434.55]

24. Secondary Outcome: Abatacept PK Parameter: Minimum Plasma Concentration at Steady State
Description: Minimum Plasma Concentration (Cmin) is the minimum observed serum drug concentration at steady state.
Time Frame: Samples were collected predose at week 8, 12, 16, 24; end of infusion at week 12; and at week 13-15 visits.
Population: All participants who received abatacept and had blood samples for assay.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | All Participants From IM101-129 Study
Number analyzed (Participants) | 113
µg/mL | 26.14 (23.10) [0.15 to 127.50]

25. Primary Outcome: Number of Participants With Vital Signs, Physical Examinations, and Electrocardiogram Findings That Were Considered to be AEs by the Investigator
Time Frame: At week 0, 2, 4; then once every 4 weeks up to 48 months; then once in every 3 months or 12 weeks to end of study (27 Dec 2010). The overall mean duration of exposure to the study drug was approximately 3 years (34.3 ± 10.7 months).
Population: All treated participants who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Number analyzed (Participants) | 13 | 178 | 26
participants
  Blood pressure increased | 2 | 27 | 12
  Blood pressure decreased | 1 | 11 | 1
  Blood pressure diastolic decreased | 0 | 7 | 0
  Blood pressure systolic increased | 0 | 3 | 2
  Weight decreased | 0 | 5 | 0
  Weight increased | 0 | 3 | 1
  Body temperature decreased | 0 | 3 | 0
  Body temperature increased | 0 | 2 | 0
  Blood pressure systolic decreased | 1 | 1 | 1
  Blood pressure diastolic increased | 0 | 1 | 0
  Electrocardiogram abnormal | 0 | 1 | 0
  Electrocardiogram ST segment depression | 0 | 1 | 0
  Electrocardiogram ST-T segment abnormal | 0 | 1 | 0
  Heart rate increased | 0 | 2 | 0
  Heart rate decreased | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg | New Participants With MTX Intolerance; Abatacept 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/13 | 50/178 | 14/26
Other Adverse Events (participants affected / at risk) | 13/13 | 176/178 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg (N=13) | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg (N=178) | New Participants With MTX Intolerance; Abatacept 10 mg/kg (N=26)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1
Radicular cyst (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Head deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pinealoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Encephalitis (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bunion operation (Surgical and medical procedures) | 0 | 1 | 0
Gastric polypectomy (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants From Phase I Study (IM101-034); Abatacept 10mg/kg (N=13) | Participants From Phase II Study(IM101-071); Abatacept 10mg/kg (N=178) | New Participants With MTX Intolerance; Abatacept 10 mg/kg (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 9 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 7 | 2
Blepharitis (Eye disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 4 | 3
Dry eye (Eye disorders) | 0 | 9 | 1
Eye discharge (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 11 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 21 | 5
Dental caries (Gastrointestinal disorders) | 0 | 21 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 10 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 3 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 7 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 2
Gastritis (Gastrointestinal disorders) | 1 | 18 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 14 | 2
Periodontitis (Gastrointestinal disorders) | 0 | 5 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 46 | 3
Toothache (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 8 | 3
Malaise (General disorders) | 1 | 8 | 1
Pyrexia (General disorders) | 1 | 11 | 4
Thirst (General disorders) | 0 | 2 | 2
Seasonal allergy (Immune system disorders) | 1 | 14 | 2
Bronchitis (Infections and infestations) | 2 | 15 | 1
Cystitis (Infections and infestations) | 4 | 11 | 0
Dermatitis infected (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 4 | 0
Gastroenteritis (Infections and infestations) | 2 | 16 | 3
Herpes simplex (Infections and infestations) | 1 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 9 | 1
Nasopharyngitis (Infections and infestations) | 8 | 103 | 12
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 5 | 0
Oral herpes (Infections and infestations) | 1 | 8 | 1
Pharyngitis (Infections and infestations) | 0 | 24 | 4
Rhinitis (Infections and infestations) | 0 | 9 | 0
Sinusitis (Infections and infestations) | 0 | 11 | 2
Tinea pedis (Infections and infestations) | 1 | 10 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 9 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 29 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 23 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 7 | 3
Blood glucose increased (Investigations) | 1 | 9 | 3
Blood pressure decreased (Investigations) | 1 | 11 | 1
Blood pressure increased (Investigations) | 2 | 27 | 12
Blood pressure systolic decreased (Investigations) | 1 | 1 | 1
Blood pressure systolic increased (Investigations) | 0 | 3 | 2
Blood urea increased (Investigations) | 1 | 6 | 0
Blood urine present (Investigations) | 1 | 14 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 9 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 15 | 1
Glucose urine present (Investigations) | 0 | 11 | 2
Lymphocyte count decreased (Investigations) | 1 | 35 | 5
Protein total decreased (Investigations) | 0 | 4 | 2
Red blood cells urine positive (Investigations) | 1 | 13 | 2
White blood cell count increased (Investigations) | 1 | 29 | 7
White blood cells urine positive (Investigations) | 3 | 18 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 22 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 12 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 8 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 9 | 3
Headache (Nervous system disorders) | 0 | 15 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 7 | 0
Sciatica (Nervous system disorders) | 1 | 3 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 20 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 21 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 28 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 29 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 15 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 15 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 2 | 13 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.